CLINICAL TRIAL: NCT05868850
Title: Study On The Application of Auricular Point Sticking Based On Holographic Theory In Chemotherapy-related Taste Alterations In Cancer Patients
Brief Title: Application of Auricular Point Sticking in Patients With Taste Alteration
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Affiliated Hospital of Jiangnan University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1415322141
Record Dates: First submitted 2023-04-24; First posted 2023-05-22 (Actual); Last update posted 2024-01-31 (Actual); Status verified 2024-01

CONDITIONS: Dysgeusia; Acupressure; Chemotherapy Effect
MeSH Terms: conditions — Dysgeusia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Routine care group (No Intervention): The control group receives routine nursing, including admission education, routine nursing of adverse reactions to chemotherapy, diet guidance for chemotherapy patients, precautions for various examinations, discharge guidance and follow-up.
- Auricular point sticking group (Experimental): Auricular point sticking therapy is performed on the basis of control group. The acupoint intervention group is established, and the research team consists of 2 graduate students, 1 graduate supervisor, 1 head nurse, 1 chief physician of traditional Chinese medicine, and 1 nursing expert. The nursing expert is responsible for the overall design of the project, and the director of traditional Chinese medicine is responsible for the selection of acupoints and the training of nurses for massage. The supervisor of graduate students and the head nurse are responsible for the overall quality control of the intervention process, while the graduate students are responsible for the preliminary and final screening of research objects, the implementation of intervention programs, the organization, coordination and recording of the entire intervention process and the collection of data.
  Interventions: Behavioral: auricular point sticking

INTERVENTIONS:
Behavioral: auricular point sticking — 1. Acupoint selection: Select Shenmen, spleen, stomach, liver, sympathetic, tongue, digestive system under the cortex, three focal, ear-back spleen.
  2. Operation: Use 75% ethanol to disinfect auricular broad skin; To be dry, use tweezers to pick up the middle of the small square tape stuck with Wang do not line seeds, align the indentation and stick well, press gently with the finger abdomen, the strength to the patient feel acid swelling, pain and heat sense and can tolerate it.
  3. Press frequency and course of treatment: it is asked to press 4 times a day, once in the morning, middle and evening before going to bed, 3-5 minutes each time, the duration of hospitalization for patients with chemotherapy is generally 3-5 days, intervention begins on the first day of chemotherapy medication, the day of discharge for patients to replace the other side of the ear acupoint, removed after 4 days of discharge. A total of 2 chemotherapy courses were treated.
  Arms: Auricular point sticking group

SUMMARY:
To explore the intervention effect of auricular point sticking on chemotherapy-induced taste alterations in cancer patients, and analyze its relationship with quality of life, nutritional status and psychology of patients.

DETAILED DESCRIPTION:
Taste alteration is a common adverse reaction in patients with chemotherapy. The incidence of taste alteration varies with chemotherapy drugs, ranging from 36% to 84%, among which platinum chemotherapeutic drugs are most likely to cause severe taste alteration. The taste alteration does not pose a serious threat to the life of patients, so it is often ignored by patients and medical staff. Dysgeusia is positively correlated with the loss of appetite, which can directly lead to the loss of appetite and insufficient intake of nutrients in patients, and even stimulate patients' anxiety, psychological pain and other negative emotions. In severe cases, it can cause malnutrition, reduce the chemotherapy compliance of cancer patients, and ultimately reduce the quality of life of patients. Therefore, for patients with platinum chemotherapy, it is necessary to pay close attention to the change of taste during chemotherapy, and apply effective nursing interventions to pay attention as soon as possible, so as to improve the quality of life of patients.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with malignant tumors diagnosed by histopathology or pathology;
2. Age ≥18 years old;
3. Patients who received platinum-based chemotherapy and completed at least one cycle of chemotherapy;
4. According to the chemotherapy-induced taste Changes Scale (CiTAS), the score of patients was ≥6;
5. Patients voluntarily participated in the treatment with good compliance and adherence.

Exclusion Criteria:

1. Patients with treatment plan adjustment or concurrent radiotherapy;
2. Patients with abnormal taste and malnutrition caused by various reasons before chemotherapy;
3. Patients with inflammation of the external ear or eczema, ulcers, chilblain in the pressing area;
4. Allergic or intolerant to adhesive stickers;
5. Those who were lost to follow-up or withdrew voluntarily;
6. Patients enrolled in other studies at the same time.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2023-06-03 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
Taste alterations | T1: Baseline. T2:2 weeks. T3: 4 weeks. T4:5 weeks.
  The Chinese version of the Chemotherapy-induced Taste Alteration Scale (CiTAS), was used to assess the patients' taste alterations. The scale has 18 items in three dimensions, namely taste alteration, unpleasant taste alteration, unpleasant symptoms and problems. The scale is a Like-5 scale with a minimum score of 18 and a maximum score of 90, with higher scores indicating more severe symptoms of taste alterations. The scale has been verified by research and has good reliability and validity.

SECONDARY OUTCOMES:
Quality of life for cancer patients | T1: Baseline. T2:2 weeks. T3: 4 weeks. T4:5 weeks. T5:8 weeks.
  With the use of the European Organization for Research on Treatment of Cancer, the most widely used guideline in clinical practice, The EORTC Quality of Life Core Questionnaire (QLQ-C30) was used to evaluate the quality of life of patients.A total of 30 items and 15 domains were included, including 5 functional domains, 9 symptom domains and 1 general health/quality of life domain. Among them, the general health status/quality of life domain was divided into 7 grades, which were calculated from 1 to 7 points according to the answer options. Other items were on a 4-point scale, and "never", "a little", "a lot" and "a lot" were scored from 1 to 4 respectively. The domain score was obtained by summing the item scores included in each domain and dividing by the number of items included, ranging from 0 to 100. A lower score indicates a better quality of life.
Anxiety and depression | T1: Baseline. T2:2 weeks. T3:4 weeks. T4:5 weeks. T5:8 weeks.
  The Chinese version of Hospital Anxiety and Depression Scale (HADS) was used to assess the anxiety and depression level of patients. There were 14 items in total, including 7 items for anxiety and 7 items for depression. Each item was scored from 0 to 3, with a minimum score of 0 and a maximum score of 42, and the higher the score, the more serious the level of anxiety and depression.
Nutritional status 1 | T1: baseline(Data were collected before the intervention). T2: 4 weeks. T3:8 weeks.
  The nutritional status of patients was evaluated according to their weight.
Nutritional status 2 | T1: baseline(Data were collected before the intervention). T2: 4 weeks. T3:8 weeks.
  The nutritional status of patients was evaluated according to their BMI.BMI= weight (in kilograms) divided by the square of height (in meters). The standard of BMI for Chinese adult residents is about 18.4, less than or equal to 18.4 is thin, 18.5 to 23.9 is normal, 24 to 27.9 is overweight, and more than or equal to 28 is obese.
Nutritional status 3 | T1: baseline(Data were collected before the intervention). T2: 4 weeks. T3:8 weeks.
  The nutritional status of patients was evaluated according weight loss rate.
Nutritional status 4 | T1: baseline(Data were collected before the intervention). T2: 4 weeks.
  The nutritional status of patients was evaluated according to their serum total protein and albumin index.

CONTACTS AND LOCATIONS:
Overall Officials: Quan Liu, Doctor, Study Chair — Affiliated Hospital of Jiangnan University
Locations (1):
- Affiliated Hospital of Jiangnan University, Wuxi, Jiangsu, China